CLINICAL TRIAL: NCT04322396
Title: Proactive Protection With Azithromycin and Hydroxychloroquine in Hospitalized Patients With COVID: A Randomized, Placebo-controlled Double-blinded Trial Evaluating Treatment With Azithromycin and Hydroxychloroquine to Patients With COVID-19
Brief Title: Proactive Protection With Azithromycin and hydroxyChloroquine in Hospitalized Patients With COVID-19
Acronym: ProPAC-COVID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recommended by the DSMB
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KronLungesyg_COVID_19_protokol
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Results first posted 2021-06-28 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Virus Diseases; Infection Viral; Corona Virus Infection
MeSH Terms: conditions — Virus Diseases; Coronavirus Infections | interventions — Azithromycin; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): This arm will receive standard care and placebo in 15 days.
  Azithromycin placebo:
  Day 1-3: 500 mg x 1 Day 4-15: 250 mg x 1
  Hydroxychloroquine placebo:
  Day 1-15: 200 mg x 2
  Interventions: Drug: Placebo oral tablet
- Intervention (Active Comparator): This arm will receive standard care and azithromycin and hydroxychloroquine in 15 days.
  Azithromycin:
  Day 1-3: 500 mg x 1 Day 4-15: 250 mg x 1
  Hydroxychloroquine:
  Day 1-15: 200 mg x 2
  Interventions: Drug: Azithromycin; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Azithromycin — Azithromycin
  Arms: Intervention
Drug: Hydroxychloroquine — Hydroxychloroquine
  Arms: Intervention
Drug: Placebo oral tablet — Placebo Azithromycin
  Arms: Control
Drug: Placebo oral tablet — Placebo Hydroxychloroquine
  Arms: Control

SUMMARY:
This study explores whether patients acutely hospitalized may have shorter hospitalization and fewer admittances at Intensive Care Units by treatment with azithromycin and hydroxychloroquine.

DETAILED DESCRIPTION:
In the ongoing coronavirus pandemic, COVID-19, that arose in Wuhan China, there is still sparse data in the course, risk of various complications, and in particular how patients who are hospitalized are best treated to ensure high survival and short hospitalization. Despite the rapid spread of the disease globally, there is no solid data yet to recommend any specific treatments, which is why symptomatic, organ supportive therapy including respiratory therapy in acute pulmonary failure is recommended. There has been reported a high incidence of bacterial super-infections in patients with COVID-19. Patients with COVID-19 also have a higher risk of dying because of septic shock. Thus, there is an urgent need for treatment that can improve the patient's chance of the shortest hospitalization possible, and treatment that can lower the risk of secondary infection and death.

This is a randomized, placebo-controlled, double-blinded multi-center trial evaluating the effect of azithromycin and hydroxychloroquine treatment in patients with COVID-19 during hospitalization. The aim of the study is to investigate whether the treatment can shorten hospitalization, reduce the risk of non-invasive ventilation, admittance to Intensive Care Units and death.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to a Danish emergency department, lung medical department or medical department
* Age >18 years
* Hospitalized <48 hours
* Positive COVID-19 test/diagnosis during the hospitalization
* Signs informed consent

Exclusion Criteria:

* If the patient uses > 5 LO2/min at time of recruitment
* Known intolerance/allergy to azithromycin or hydroxychloroquine or hypersensitivity to quinine or 4-aminoquinolinderivates
* Pregnancy
* Breastfeeding
* Neurogenic hearing loss
* Psoriasis
* Retinopathy
* Maculopathy
* Changes in vision field
* Severe liver disease other than amoebiases
* Severe gastrointestinal, neurological or haematological disorders
* eGFR < 45 ml/min/1.73m2
* Clinically significant cardiac conduction disorders/arrhythmias or prolonged QTc interval
* Myasthenia Gravis
* Uses Digoxin
* Glucose-6-phosphate dehydrogenase deficiency
* Porphyria
* Hypoglycemia at any time since hospitalization
* Severe mental illness which significantly impedes cooperation
* Severe linguistic problems that significantly impedes cooperation
* Treatment with sickle alkaloids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Denmark (8):
  - Aalborg Sygehus, Aalborg
  - Bispebjerg Hospital, Copenhagen
  - Herlev-Gentofte Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen
  - Nordsjællands Hospital, Hillerød
  - Odense Universitetshospital, Odense
  - Roskilde Sygehus, Roskilde
  - Slagelse Sygehus, Slagelse

REFERENCES:
- [Derived] Sivapalan P, Ulrik CS, Lappere TS, Eklof JV, Shaker SB, Bodtger UCS, Browatzki A, Meyer CN, Weinreich UM, Laursen CB, Biering-Sorensen T, Knop FK, Lundgren JD, Jensen JS. Proactive prophylaxis with azithromycin and hydroxychloroquine in hospitalized patients with COVID-19 (ProPAC-COVID): a statistical analysis plan. Trials. 2020 Oct 20;21(1):867. doi: 10.1186/s13063-020-04795-0. PMID 33081817
- [Derived] Sivapalan P, Ulrik CS, Bojesen RD, Lapperre TS, Eklof JV, Hakansson KEJ, Browatzki A, Tidemansen C, Wilcke JT, Janner J, Gottlieb V, Meteran H, Porsbjerg C, Madsen BL, Moberg M, Pedersen L, Benfield TL, Lundgren JD, Knop FK, Biering-Sorensen T, Ghanizada M, Sonne TP, Bodtger UCS, Jensen SG, Rasmussen DB, Brondum E, Tupper OD, Sorensen SW, Alstrup G, Laursen CB, Moller UW, Sverrild A, Jensen JS. Proactive Prophylaxis With Azithromycin and HydroxyChloroquine in Hospitalised Patients With COVID-19 (ProPAC-COVID): A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 10;21(1):513. doi: 10.1186/s13063-020-04409-9. PMID 32522282

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: This arm will receive standard care and placebo in 15 days.
  Placebo oral tablet: Placebo Azithromycin
  Placebo oral tablet: Placebo Hydroxychloroquine
- Intervention: This arm will receive standard care and azithromycin and hydroxychloroquine in 15 days.
  Azithromycin: Azithromycin
  Hydroxychloroquine: Hydroxychloroquine
Period: Overall Study
Arm/Group | Control | Intervention
Started | 56 | 61
Completed | 56 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 56 | 61 | 117
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [52 to 74] | 68 [52 to 80] | 65 [52 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 29 | 36 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Caucasian | 45 | 53 | 98
  Race/ethnicity: African | 1 | 0 | 1
  Race/ethnicity: Asian | 6 | 6 | 12
  Race/ethnicity: Unknown/other | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 56 | 61 | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Alive and Discharged From Hospital Within 14 Days
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
days | 9 [7 to 10] | 9 [3 to 11]

2. Secondary Outcome: Categorization of Hospitalization Status
Description: The patient will be categorized into one of the following 8 categories depending on status of their hospitalization:
  1. Dead (yes/no)
  2. Hospitalized and receiving mechanical ventilation or ExtraCorporalMembraneOxygenation (ECMO) (yes/no)
  3. Hospitalized and receiving Non-invasive ventilation or "high-flow oxygen device" (yes/no)
  4. Hospitalized and given oxygen supplements different from (2) and (3) (yes/no)
  5. Hospitalized and without oxygen treatment, but receiving other treatment (both related to COVID-19 or other) (yes/no)
  6. Hospitalized for observation (yes/no)
  7. Discharged from hospital with restriction of activity level (yes/no)
  8. Discharged from hospital without any restrictions of activity level (yes/no)
  Only one category can be "yes".
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
Participants
  Dead | 2 | 1
  Hospitalized and receiving mechanical ventilation or ExtraCorporalMembraneOxygenation (ECMO) | 1 | 3
  Hospitalized and receiving Non-invasive ventilation or "high-flow oxygen device" | 0 | 1
  Hospitalized and given oxygen supplements different from (2) and (3) | 2 | 2
  Hospitalized and without oxygen, but receiving other treatment (both related to COVID-19 or other) | 2 | 1
  Hospitalized for observation | 0 | 1
  Discharged from hospital with restriction of activity level | 27 | 26
  Discharged from hospital without any restrictions of activity level | 22 | 26

3. Secondary Outcome: Length of Stay in ICU
Description: Length of stay in intensive care unit.
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
days | 11 [4 to 14] | 14 [9.5 to 14]

4. Secondary Outcome: Number of Participants on Non-invasive Ventilation (NIV) During Hospitalization
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
Participants | 1 | 3

5. Secondary Outcome: Mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
Participants | 2 | 1

6. Secondary Outcome: Length of Hospitalization
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
days | 4 [3 to 6] | 4 [2 to 8]

7. Secondary Outcome: Days Alive and Discharged From Hospital
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
days | 26 [23 to 27] | 26 [21 to 28]

8. Secondary Outcome: Mortality
Time Frame: 90 days
Reporting Status: Not Posted

9. Secondary Outcome: Mortality
Time Frame: 365 days
Reporting Status: Not Posted

10. Secondary Outcome: Number of Readmissions (All Causes)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
Participants | 6 | 9

11. Secondary Outcome: Number of Days Using Non-invasive Ventilation (NIV)
Description: Number of days using non-invasive ventilation (NIV) if on NIV during hospitalization.
Time Frame: 14 days
Population: The Overall Number of Participants Analyzed represents the number of participants with available data.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 1 | 3
days | 9.0 [NA to NA] — Only 1 patient on NIV in this group. | 6.7 [-9.1 to 22.4]

12. Secondary Outcome: Change in Patient's Oxygen Partial Pressure
Description: PaO2 measured in arterial puncture at baseline and 4 days.
Time Frame: 4 days
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
mmHg | -0.2 [-8.3 to 7.8] | -3.0 [-9.8 to 3.9]

13. Secondary Outcome: Change in Patient's Carbondioxide Partial Pressure
Description: PaCO2 measured in arterial puncture at baseline and 4 days.
Time Frame: 4 days
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
mmHg | 1.4 [-0.4 to 3.3] | -3.0 [-9.8 to 3.9]

14. Secondary Outcome: Change of pH in Blood
Description: pH measured in arterial puncture at baseline and 4 days.
Time Frame: 4 days
Measure: Mean (95% Confidence Interval); unit: pH
Arm/Group | Control | Intervention
Number analyzed (Participants) | 56 | 61
pH | 0.0 [-0.02 to 0.01] | 0.0 [-0.03 to 0.01]

15. Secondary Outcome: Time for no Oxygen Supplement (or Regular Oxygen Supplement "LTOT")
Description: Time for no oxygen supplement (or regular oxygen supplement "LTOT") if on oxygen during admission.
Time Frame: 14 days
Population: The Overall Number of Participants Analyzed represents the number of participants with available data
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Control | Intervention
Number analyzed (Participants) | 27 | 25
hours | 72 [39.75 to 96] | 72 [24 to 192]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the period beginning when the patient received their first dose of trial medication up to and including day 15. All-Cause Mortality was assessed up to 30 days.
Description: A serious adverse event (SAE) was defined as an event or adverse event that, regardless of dose, was life-threatening, resulted in significant or persistent disability or incapacity, or led to a congenital anomaly or malformation.
  Because comorbidities and mortality are common in this patient group, prolonged admission, re-admission, non-invasive ventilation, invasive respiratory treatment and death were not considered SAEs.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 2/56 | 1/61
Serious Adverse Events (participants affected / at risk) | 2/56 | 0/61
Other Adverse Events (participants affected / at risk) | 25/56 | 31/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=56) | Intervention (N=61)
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Hearing loss (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0
Seizure (Nervous system disorders) | 0 | 0
Stroke (Nervous system disorders) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=56) | Intervention (N=61)
Prolonged QTc (Cardiac disorders) | 7 | 4
Chest pain (Cardiac disorders) | 4 | 3
Hypoglycaemia (Endocrine disorders) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 12
Vomiting (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 6 | 11
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Headache (Nervous system disorders) | 5 | 3
Photophobia (Nervous system disorders) | 0 | 0
Dizziness (Nervous system disorders) | 3 | 10
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Itching/Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Bleeding (Vascular disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Early termination based on recommendations from the DSMB leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT04322396/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT04322396/SAP_001.pdf